CLINICAL TRIAL: NCT00956917
Title: Comparison of Impedance Components and Estimated Body Composition Variables Determined by Using Bioelectrical Impedance Devices Manufactured by Akern SRL and RJL Systems
Brief Title: Comparison Study for Bioelectrical Impedance Device to Measure Human Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akern USA LLC (Industry)
Responsible Party: Michaeal G. Singer, Akern USA LLC
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: EFG001
Record Dates: First submitted 2009-08-08; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Body Composition Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Akern EFG (Active Comparator)
  Interventions: Device: Akern USA EFG
- RJL device (Active Comparator)
  Interventions: Device: RJL Impedance analyzer

INTERVENTIONS:
Device: Akern USA EFG — Impedance measurement device
  Arms: Akern EFG
Device: RJL Impedance analyzer — Impedance analyzer
  Arms: RJL device

SUMMARY:
The purpose of this study is to determine if the ElectroFluidGraph(tm) (EFG) impedance analyzer is comparable to a predicate device in measuring human body composition.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the ElectroFluidGraph(tm) (EFG) impedance analyzer is comparable to a predicate device in measuring human body composition under normal patient conditions. Specifically, the goal of this study is to compare impedance measurements (R and Xc) determined by using each bioelectrical impedance device and the estimated body compositional estimates [total body water (TBW); fat-free mass (FFM); and fat mass (FM)] calculated by using the same prediction equation (models) as the predicate device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* None

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Resistance (R) - (ohms) | 5 minutes

SECONDARY OUTCOMES:
Fat Free Mass (FFM) | 5 minutes
Total Body Water (TBW) | 5 minutes
Extra Cellular Water | 5 minutes
Fat Mass (FM) | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gatteschi, MD, Principal Investigator
Locations (1):
- Laboratorio, FIGC, Settore Tecnico Coverciano, D'Annunzio, Florence, Italy